CLINICAL TRIAL: NCT06390826
Title: MATCH Treatment Subprotocol V: Phase II Study of Sunitinib in Patients With Tumors With cKIT Mutations (Excluding GIST, Renal Cell Carcinoma or Pancreatic Neuorendocrine Tumor)
Brief Title: Testing Sunitinib as Potentially Targeted Treatment in Cancers With cKIT Genetic Changes (MATCH - Subprotocol V)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01135; NCI-2024-01135 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-V (Other: ECOG-ACRIN Cancer Research Group); EAY131-V (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-27; First posted 2024-04-30 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (sunitinib) (Experimental): Patients receive sunitinib 50 mg PO QD on days 1-28 of each cycle. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo ECHO or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Radionuclide Imaging; Drug: Sunitinib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Radionuclide Imaging — Undergo nuclear study
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Drug: Sunitinib — Given PO

SUMMARY:
This phase II MATCH treatment trial tests how well sunitinib in treating patients with cancer that has certain genetic changes. Sunitinib is in a class of medications called kinase inhibitors. It is used in patients whose cancer has a certain mutation (change) in the cKIT gene. It works by blocking the action of mutated cKIT that signals cancer cells to multiply. This helps to stop or slow the spread of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive sunitinib 50 mg orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 42 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study, as well as during follow-up as clinically necessary. Patients also undergo echocardiography (ECHO) or nuclear study throughout the trial as clinically necessary. Patients undergo biopsies and blood sample collection on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria of MATCH Master Protocol at the time of registration to treatment step (Step 1, 3, 5, 7)
* Patients must have a somatic cKIT mutation in exon 9, 11, 13 or 14, excluding exon 17 or 18 mutations, activating PDGFRA or PDGFRB variants and fusions, or another aberration, as identified via the MATCH Master Protocol

  * Actionable mutations of interest (aMOIs)for information on the inclusion and exclusion mutations, along with the corresponding levels of evidence (LOE)
* Total bilirubin must be within normal institutional limits
* Creatinine must be within normal institutional limits. OR Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Serum calcium must be =< 12.0 mg/dL
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with known left ventricular dysfunction must have ECHO or a nuclear study (multigated acquisition scan [MUGA] or first pass) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible.

  * The following groups of patients are eligible provided they have New York Heart Association class II cardiac function on baseline ECHO/nuclear study:

    * Patients with a history of class II heart failure who are asymptomatic on treatment
    * Patients with prior anthracycline exposure
    * Patients who have received central thoracic radiation that included the heart in the radiotherapy port NOTE: Pre-treatment LVEF determination in patients without known left ventricular dysfunction (or per Section 2.1.5.1) is NOT otherwise required
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
  * History of pulmonary embolism within the past 12 months
* Patients must not have known hypersensitivity or excess toxicity from sunitinib or compounds of similar chemical composition or biologic effect. This list includes, but is not limited to, patients with significant cardiac or hepatic toxicity from multikinase inhibitors with similar kinase inhibitory profiles (sorafenib, regorafenib, pazopanib)

  * Questions regarding a significant intolerance to a prior therapy should be directed to the sub-protocol principal investigator (PI)
* Patients must not have had prior therapy with sunitinib
* Patients must not have planned ongoing administration of STRONG and MODERATE CYP3A4 inhibitors or inducers. The reference list of cytochrome p450 (CYP) isozymes and classification of strong, moderate, and weak interactions is available through the FDA website

  * Strong CYP3A4 inhibitors are not permitted within 7 days before dosing and should be avoided throughout the study
  * Strong CYP3A4 inducers are not permitted within 12 days before dosing and should be avoided throughout the study
* Patients must not have gastrointestinal stromal tumor (GIST), renal cell carcinoma, or pancreatic neuroendocrine tumor
* Patients must not have a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4 grade 3 hemorrhage within 4 weeks of starting study treatment
* Patients must not have hypertension that cannot be controlled by medications (> 140/90 mmHg despite optimal medical therapy)
* Patients must not have pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Participants may not have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting sunitinib
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients who require therapeutic doses of coumarin derivative anticoagulants such as warfarin are excluded, although doses up to 2 mg daily are permitted for prophylaxis of thrombosis NOTE: Low molecular weight heparin is permitted provided that the patient's prothrombin time (PT) international normalized ratio (INR) is < 1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian T Gien, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol V was activated on August 12, 2015. A total of 10 patients were enrolled between November 1, 2016 and May 21, 2020. Four patients were enrolled on the basis of the results from the NCI-MATCH assay and 6 on the basis of the outside assay results.
Pre-assignment Details: Eligible patients for arm-V must have a somatic cKIT mutation in exon 9, 11, 13 or 14, excluding exon 17 or 18 mutations, activating PDGFRA or PDGFRB variants and fusions, or another aberration as identified in the protocol. The mutation status was determined by an NCI-MATCH approved laboratory for 6 patients in this arm, these cases had to be confirmed to be used in primary analysis.
Period: Overall Study
Arm/Group | Treatment (Sunitinib)
Started | 10
Started Protocol Therapy | 9
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 9
Completed | 0
Not Completed | 10
Not completed — Never Start Protocol Therapy | 1
Not completed — Adverse Event | 1
Not completed — Disease Progression | 8

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Sunitinib)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 62 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.* For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)
Time Frame: Tumor assessments occurred at baseline, then every 3 months if patient is < 2 years from study entry, and every 6 months thereafter until disease progression, up to 3 years post registration
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Sunitinib)
Number analyzed (Participants) | 9
percentage of participants | 22.2 [4.1 to 55]

2. Secondary Outcome: 6-month Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Sunitinib)
Number analyzed (Participants) | 9
percentage of participants | 33.3 [15.4 to 72.4]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Sunitinib)
Number analyzed (Participants) | 9
months | 4.2 [2.9 to 8.5]

ADVERSE EVENTS:
Time Frame: Assessed every 42 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Nine patients were included in the toxicity analysis (excluding one who did not receive treatment).
Arm/Group | Treatment (Sunitinib)
All-Cause Mortality (participants affected / at risk) | 7/10
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib) (N=9)
Fatigue (General disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib) (N=9)
Anemia (Blood and lymphatic system disorders) | 3
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Chills (General disorders) | 1
Edema face (General disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Localized edema (General disorders) | 1
Pain (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 5
White blood cell decreased (Investigations) | 4
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 4
Irregular menstruation (Reproductive system and breast disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT06390826/Prot_000.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT06390826/ICF_001.pdf